CLINICAL TRIAL: NCT01457404
Title: Integrated Cognitive Behavioral Therapy for Co-Occurring PTSD and Substance Use Disorders
Brief Title: Integrated Cognitive Behavioral Therapy (ICBT) for Posttraumatic Stress Disorder (PTSD) and Substance Use Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Brown University (Other); Providence VA Medical Center (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark McGovern, Associate Professor of Psychiatry and of Community and Family Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA030102 (NIH); 5R01DA030102 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-24 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Stress Disorder, Post-Traumatic; Substance-Related Disorders
Keywords: integrated cognitive behavioral therapy; cognitive behavioral therapy; addiction; posttraumatic stress disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Cognitive Behavioral Therapy (Experimental): Integrated Cognitive Behavioral Therapy (ICBT) is a non-exposure based, manual-guided individual or group therapy. ICBT consists of 3 learning and skill components designed to improve PTSD symptoms and substance use: 1) Patient education about PTSD and its relation to substance use and treatment; 2) Mindful relaxation: A behavioral anxiety reduction skill including centering and breathing techniques; and 3) Cognitive restructuring/flexible thinking: A cognitive approach and functional analysis of the link among emotions, cognitives and situations.
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy
- Treatment-as-usual (Active Comparator): Treatment-as-usual (TAU) is the typical outpatient treatment that patients would receive ordinarily at the PVAMC Substance Abuse Treatment Program (SATP) or PTSD Clinic.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Integrated Cognitive Behavioral Therapy — Individual or group ICBT, approx. 12 sessions, one session per week
  Other Names: ICBT; CBT for PTSD; CBT
  Arms: Integrated Cognitive Behavioral Therapy
Behavioral: Treatment-as-usual — Individual or group therapy as usual within the SATP or PTSD clinics at the PVAMC
  Other Names: TAU
  Arms: Treatment-as-usual

SUMMARY:
The purpose of this study is to assess the safety and practicality, feasibility and efficacy of ICBT for co-occurring PTSD and substance use disorders within the OEF/OIF/OND Veterans population, as delivered by routine clinicians at the Veterans Affairs.

DETAILED DESCRIPTION:
The proposed research will evaluate the safety and practicality, feasibility, and efficacy of a relatively simple, manual guided integrated cognitive behavioral therapy (ICBT). ICBT (a revised edition of what was formerly called cognitive behavioral therapy for posttraumatic stress disorder [CBT for PTSD]) has been designed and developed for delivery by counselors employed in community addiction treatment programs and offered in conjunction with standard community addiction treatment. The investigators have completed a Stage I Safety & Practicality Study, Feasibility Study and Pilot Randomized Controlled Study (comparing ICBT versus a control condition) in community addiction treatment and for all studies found that ICBT was safe and effective in reducing PTSD symptoms, improving retention, and in reducing substance use. The present study proposes to conduct a Stage I study of ICBT among Operation Enduring Freedom (OEF) Operation Iraqi Freedom (OIF) and Operation New Dawn (OND) Veterans within the Veterans Affairs treatment setting. The investigators will modify the existing ICBT for testing in a VA setting, and use a combined individual and group modality.

There are 3 specific aims for this study, and hypotheses for each aim:

Aim 1: To test the feasibility of ICBT with OEF/OIF/OND Veterans diagnosed with PTSD and substance use disorders, and assess substance use and PTSD outcomes at 3- and 6-month follow-up (Stage I Phase I: Safety and practicality testing; Feasibility Study).

* This aim is to test the effect of ICBT on symptoms of PTSD and substance use disorders among returning OEF/OIF/OND Veterans seen in a VA clinic. ICBT will be tested with 16 Veterans who meet criteria for both PTSD and substance use disorder at the PTSD or SATP clinics. The investigators propose that ICBT will result in significant reductions in PTSD and substance use severity from baseline to follow-up assessment.
* Hypothesis 1: Participants receiving ICBT will have significant reductions in PTSD symptom severity as assessed by their Clinician Administered PTSD Scale (CAPS) score from baseline to a 6-month follow-up assessment.
* Hypothesis 2: Participants receiving ICBT will have significant reductions in substance use as assessed by their Addiction Severity Index (ASI) drug and alcohol severity composite scores from baseline to a 6-month follow-up assessment.

Aim 2: To revise the ICBT materials and protocol based on Stage I Phase I findings (Stage I Phase II).

-Based on experience and lessons learned in Stage I Phase I, the investigators will refine and improve the ICBT approach and study methods for teh Stage I Phase III randomized pilot trial.

Aim 3: To conduct a randomized controlled pilot trial comparing ICBT plus standard Substance Abuse Treatment Program (SATP) or PTSD care versus standard SATP or PTSD care alone, with OEF/OIF/OND Veterans diagnosed with PTSD and substance use disorders, and assess substance use and PTSD outcomes at post treatment and 3-month post treatment follow-up (Stage I Phase III: Randomized Pilot Trial).

* The efficacy of ICBT will be tested among 64 Veterans who screen positive for both disorders and are randomly assigned to either ICBT or standard treatment.
* Hypothesis 1: Participants receiving ICBT plus standard care will have greater reductions in PTSD symptoms, as assessed by their CAPS score from baseline to follow-up, than participants receiving standard care alone.
* Hypothesis 2: Participants receiving ICBT plus standard care will have greater reductions in substance use, as assessed by their ASI drug and alcohol severity composite scores from baseline to follow-up, as compared to participants receiving standard care alone.

Potential subjects will be receiving PTSD or substance use treatment services at the Providence Veterans Affairs Medical Center (PVAMC), and will be referred by clinicians in these respective clinics for participation in the study. Patients will be approached by the clinic staff about potential interest in the study. If they wish to learn more about the study, the research coordinator (an on-site employee) is contacted, a suitable time arranged, and the patient is engaged in the process of informed consent.

If consent is granted, the subjects completes the baseline assessment. The baseline assessment consists of measures gathered via interview by a member of the research team, self-administered surveys completed directly by the subject, and review of the subject's medical record to extract demographic, substance use, and treatment history information, as well as chart diagnoses.

The interview portion of the assessment consists of:

* Standardized interviews designed to assess PTSD and Axis I DSM-IV substance use disorders: Clinician Administered PTSD Scale (CAPS) and the Structured Clinical Interview for DSM-IV-TR, Patient Edition (SCID-I/P) Section E.
* A urine screen and breathalyzer to test for alcohol and other drugs.
* Standardized follow-back method for gathering data on recent alcohol and drug use: Time-line Follow-back Calendar (TLFB).

The self-administered portion of the assessment consists of measures designed to assess:

* Alcohol and drug use, as well as associated problems in other life areas such as medical, employment, legal, social, and psychiatric: Addiction Severity Index (ASI).
* Depression: Patient Health Questionnaire-9 (PHQ-9).

If the subject continues to meet criteria for PTSD (i.e. the CAPS interview confirms diagnosis of DSM-IV PTSD, with symptom severity at 44 or higher), he or she is eligible to participate. For Stage I Phase I, the patient would receive the ICBT therapy. For Stage I Phase III, the patient would be randomized to receive either the ICBT therapy plus standard treatment, or standard treatment only.

Research assessments are then also conducted at three months and six months post baseline assessment. This follow-up assessment will consist of the same measures administered at baseline, with the exception of the SCID interview.

The investigators plan to enroll approximately 16 subjects in the Stage I Phase I and to randomize approximately 64 subjects in the Stage I Phase III of the study. The subject outcome and program experiences with the protocol will be used in planning the subsequent federal grant application for a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. OEF/OIF/OND Veteran status;
2. Diagnosis of PTSD confirmed by the Clinician Administered PTSD Scale (CAPS) with a total symptom score of 44 or more;
3. Diagnosis of a substance use disorder (abuse or dependence) and confirmed by the Structured Clinical Interview of DSM-IV Section E (SCID-E);
4. Willing and able to provide informed consent;

Exclusion Criteria:

1. Acute psychotic symptoms (however, persons with a psychotic disorder are eligible if their symptoms are stable and they are well connected with appropriate mental health services);
2. Psychiatric hospitalization or suicide attempt in the past month (however, if the hospitalization or attempt was directly related substance intoxication or detoxification and ther person is currently stable, they are eligible);
3. Medical or legal situations are unstable such that ability to participate in the full duration of the study seems unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Decrease from baseline in Clinician Administered PTSD Scale (CAPS) score (PTSD symptom severity) at 3-months and at 6-months | Baseline, post-treatment, 3 months post treatment

SECONDARY OUTCOMES:
Reduction from baseline in substance use severity (Addiction Severity Index [ASI]) at 3-months and at 6-months | Baseline, post treatment, 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. McGovern, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Providence Veterans Affairs Medical Center (PVAMC), Providence, Rhode Island, United States